CLINICAL TRIAL: NCT05223153
Title: Assessment of Macular Microvascular Changes Following Amblyopia Treatment in Children With Anisometropic Amblyopia Using Optical Coherence Tomography Angiography
Brief Title: OCT-A and Amblyopia
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sahar T A Abdelaziz, Assistant Professor, Minia University
Other Study IDs: Ophthalomlogy department
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amblyopic eye group
  Interventions: Diagnostic Test: Optical Coherence tomography angiography
- Sound eye group
  Interventions: Diagnostic Test: Optical Coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence tomography angiography — Measurement retinal vessel density in the superficial and deep capillary plexuses using OCTA in children with anisometropic amblyopia

SUMMARY:
Detect changes in retinal vessel density in the superficial and deep capillary plexuses using OCTA in children with anisometropic amblyopia

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral anisometropia.
2. Refractive error less than -6.00 D and +4.00 D.
3. Age less than 12 years.
4. No previous amblyopia treatments

Exclusion Criteria:

1. High refractive error. 2. Bilateral amblyopia. 3. Age more than 12 years.

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with unilateral anisometropic amblyopia without previous treatment with glasses or patches
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in retinal vessel density | 3 months
  Detect changes in retinal vessel density in the superficial and deep capillary plexuses using OCTA in children with anisometropic amblyopia and effect of treatment on the retinal vessel density

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AttaAllah HR, Abdelaziz STA, Mohamed AAM, Ibrahiem MFK. Assessment of macular microvascular changes in children following treatment of anisometropic myopic amblyopia using optical coherence tomography angiography. Graefes Arch Clin Exp Ophthalmol. 2023 Sep;261(9):2689-2699. doi: 10.1007/s00417-023-06055-8. Epub 2023 Apr 13. PMID 37052667